CLINICAL TRIAL: NCT00409604
Title: Clinical Evaluation of Pacing During the Onset of Revascularization / Feasibility Study
Brief Title: PROTECT : Pacing to Protect Heart for Damage From Blocked Heart Vessel and From Re-opening Blocked Vessel(s)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guidant Corporation (Industry)
Responsible Party: Racho Strauven, Guidant Europe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS1017-001
Record Dates: First submitted 2006-12-08; First posted 2006-12-11 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Acute Myocardial Infarction

ARMS (2):
- 1 (Experimental): Standard PCI procedure + pacing post conditioning
  Interventions: Device: Temporary RV VVI pacing
- 2 (No Intervention): Standard PCI procedure

INTERVENTIONS:
Device: Temporary RV VVI pacing — temporary pacing at the onset of revascularisation
  Arms: 1

SUMMARY:
To determine whether the application of ventricular pacing can protect the human heart from damage resulting from a myocardial infarction

DETAILED DESCRIPTION:
To determine whether the application of ventricular pacing can protect the human heart from damage resulting from a myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute myocardial infarction, requiring PCI within 2 to 6 hours following symptoms
* Total occlusion of a coronary artery with reference vessel diameter >or= 3mm

Exclusion Criteria:

* Thrombolitics
* Severe bradycardia requiring cardiac pacing
* Previous PCI or CABG
* Recent stroke or CV surgery
* Recent major surgery or trauma
* Clinical and hemodynamic unstability
* Implanted CRM device
* Evidence of previous MI
* Diabetes using rosiglitazone or other fibrates
* Permanent AF
* Mechanical tricuspid valve
* Pregnancy
* Exclusion for MRI
* Incapability of participating in exercise test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Infarct size (area under the curve of creatine kinase) at baseline compared with MRI at 4 months and at 12 months | 4 & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: JOhannes Waltenberger, Prof.Dr., Principal Investigator — University Hospital of Maastricht (azM), P. Debyelaan 25, 6202 AZ Maastricht, The Netherlands
Locations (1):
- University Hospital of Maastricht (azM), Maastricht, Netherlands

REFERENCES:
- [Derived] Waltenberger J, Gelissen M, Bekkers SC, Vainer J, van Ommen V, Eerens F, Ruiters A, Holthuijsen A, Cuesta P, Strauven R, Mokelke E, Gorgels A, Prinzen FW. Clinical pacing post-conditioning during revascularization after AMI. JACC Cardiovasc Imaging. 2014 Jun;7(6):620-6. doi: 10.1016/j.jcmg.2014.01.017. PMID 24925330